CLINICAL TRIAL: NCT02950909
Title: Effect of Therapeutic Exercise on the Activation of the Neck Extensors in People With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moisés Giménez Costa (Other)
Responsible Party: Sponsor-Investigator, Moisés Giménez Costa, Associated professor, University of Valencia
Organization: University of Valencia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1472552616890
Record Dates: First submitted 2016-10-25; First posted 2016-11-01 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Neck Pain
Keywords: Therapeutic exercise; Chronic pain; Neck extensors
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emphasized exercise group (Experimental): Patients in the emphasized exercise group performed exercises emphasizing the deep cervical extensor muscles applying a resistance at the level of the vertebral arch of C4 either therapeutically with the therapist's fingers or as a home exercise with the aid of a towel or belt. These exercises were performed in sitting and standing in front of a table propped up on both forearms. In the latter position, a dynamic exercise was added moving the head from maximal flexion to maximal extension keeping the gaze fixed at an object lying between both elbows hoping to activate more the extensors in the lower cervical spine.
  Interventions: Procedure: Static exercise for emphasized neck extensors; Procedure: Dynamic exercise for emphasized neck extensors
- General exercise group (Experimental): Patients in the general exercise group performed exercises targeting all cervical extensor muscles including the superficial ones applying resistance at the head pushing against a wall or the therapist's hand or as a home exercise with the aid of a towel. As in the other group, these exercises were performed in sitting and standing in front of a table propped up on both forearms. In the latter position, the same dynamic exercise was added as in the other group with the only difference that the gaze was fixed at an object lying between both hands hoping to activate all cervical extensors
  Interventions: Procedure: Static exercise for general neck extensors; Procedure: Dynamic exercise for general neck extensors

INTERVENTIONS:
Procedure: Static exercise for emphasized neck extensors — Emphasized activation of the deep neck extensors was searched for applying a localized resistance with the thumb and index finger at the level of the vertebral arch of C4 while pushing into flexion in a ventral-cranial direction, approximately parallel to the surface of the zygapophyseal joint, asking the patient to resist maximally during 6 seconds in sitting position
  Arms: Emphasized exercise group
Procedure: Dynamic exercise for emphasized neck extensors — The patient was asked to fix his gaze at an object lying between both elbows hoping to in order to emphasize extension in the lower cervical spine and consequently activation of the extensors in this region.
  Arms: Emphasized exercise group
Procedure: Static exercise for general neck extensors — Emphasized activation of all neck extensors was searched for applying the resistance with the therapist's hand or a wall respectively a towel at the occiput in sitting position
  Arms: General exercise group
Procedure: Dynamic exercise for general neck extensors — . The patient was asked to fix his gaze at an object lying between both hands. Extension consequently occurred in the entire cervical spine.
  Arms: General exercise group

SUMMARY:
The primary aim of this study therefore is to investigate the effects on pain and disability of an emphasized exercise program targeting the deep neck extensor semispinalis cervicis and a general exercise program for all neck extensor muscles in patients with chronic neck pain. As a secondary aim , pain intensity (VAS), cervical ROM, pressure pain threshold (PPT), cervical and thoracic posture and self-perceived benefit of treatment (GROC) were measured. The investigators hypothesized that both exercise programs would have similar effects on pain alleviation and pain related disability, but that the emphasized exercise program for the deep semispinalis cervicis would improve its activation more compared to the general exercise program. The results of this study will be relevant for designing effective rehabilitation/training programs for patients with chronic neck pain.

DETAILED DESCRIPTION:
An independent group, repeated-measures study design was adopted to investigate the immediate effect of two different kinds of intervention: Emphasized exercises targeting the deep cervical extensors and general exercises targeting all neck extensors. Subjects were randomized into two exercise groups: the emphasized exercise group in which patients performed muscle contractions against resistance directly at the neck and the general exercise group in which the resistance was applied at the head. Sealed opaque envelopes were used to conceal allocation.

Exercise regimes was of 6-weeks duration and started within one week of the initial assessment. All subjects received personal instruction and supervision by one experienced physiotherapist, once a week, for the duration of the whole program.

Subjects received an exercise diary and were requested to practice their respective regime twice per day for the six-week duration of the trial, without provoking neck pain and with attention to correct performance of the exercises. Exercises at home occurred for a period of no longer than 15 to 20 minutes twice per day. Subjects were asked not to seek other interventions for neck pain during the duration of the study, although usual medication was not withheld.

All patients performed two static exercises and one dynamic exercise. The only difference between both groups was the location of the resistance, which was in the lower cervical spine approximately at level C4 for the emphasized exercise group and at the occiput for the general exercise group.

1. Patients in the emphasized exercise group performed exercises emphasizing the deep cervical extensor muscles applying a resistance at the level of the vertebral arch of C4 either therapeutically with the therapist's fingers or as a home exercise with the aid of a towel or belt. These exercises were performed in sitting and standing in front of a table propped up on both forearms. In the latter position, a dynamic exercise was added moving the head from maximal flexion to maximal extension keeping the gaze fixed at an object lying between both elbows hoping to activate more the extensors in the lower cervical spine.
2. Patients in the general exercise group performed exercises targeting all cervical extensor muscles including the superficial ones applying resistance at the head pushing against a wall or the therapist's hand or as a home exercise with the aid of a towel. As in the other group, these exercises were performed in sitting and standing in front of a table propped up on both forearms. In the latter position, the same dynamic exercise was added as in the other group with the only difference that the gaze was fixed at an object lying between both hands hoping to activate all cervical extensors.

The dosage for both exercise regimes required maximal muscle activation of the patient because it was shown that at this dosage the emphasized exercise results in muscle activation of about 20% to 25% MVC (Maximum Voluntary Contraction) and the general exercise of about 50% MVC (Schomacher et al., 2015). Patients were asked therefore to perform the exercises at their individual maximal force for a short time without provoking any pain neither during nor after the exercise. That is, submaximal effort without evoking pain during and after the exercises was used.

All exercises were repeated each for 3 sets with a break of 1-2 minutes between the sets. The two static exercises consisted of 6 repetitions of 6 seconds hold in each position with 6 seconds rest between each contraction. The dynamic exercise was performed with 6 repetitions through the whole range of motion with 2-3 seconds for each repetition without any rest between the repetitions. A break between the repetitions was added if necessary to avoid pain (Table 1). Patients repeated the exercise session one time per week under supervision of a physiotherapist, during 6 weeks. In addition, patients performed the exercise session twice per day seven days per week at home. Each exercise session lasted about 20 - 25 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate pain intensity between 3 and 5 from 10 Visual Analogue Scale)to avoid exacerbation of pain with the neck exercises;.
* Poor performance in the neck extensor resistance test as described by Lee et al. (Lee et al., 2005) and Parazza et al. (Parazza et al., 2014) of less than 250 seconds , which justify the application of an exercise program in the neck extensors.

Exclusion Criteria:

* neurological signs in the upper limb
* any contraindication for EMG like known risk of having infection following clinical needle insertion, coagulation disorders or medications affecting coagulation like aspirin
* pregnancy
* if they had participated in a neck exercise program in the past 12 months or had cervical spine surgery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 3 months
  Variation in the Neck Disability Index scale

SECONDARY OUTCOMES:
Neck pain intensity (Visual Analogue Scale) | 6 months
  Variation of 2 or more in the Scale
Range of motion | 7 weeks
  Measurements in goniometric degrees for neck flexion, extension, sidebending (left and right) and rotation (left and right)
Pressure pain threshold | 7 weeks
  Measurement using a digital algometer positioned over the zygapophyseal joints of C2 and C5 on the most painful side, or on the right side when both sides were equally painful. In addition, a remote PPT site on the right tibialis anterior
Global Rating of Change scale | 7 weeks
  Modification of the perceived pain and disability status with the questionary

CONTACTS AND LOCATIONS:
Overall Officials: Moises Giménez-Costa, Investigator, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT02950909/ICF_000.pdf